CLINICAL TRIAL: NCT02195830
Title: Bedside Ultrasound of Inferior Vena Cava Collapsibility in Emergency Department Patients Presenting With Severe Sepsis and Septic Shock
Brief Title: Inferior Vena Cava Collapsibility Index in Severe Sepsis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Teesside University (Other)
Responsible Party: Principal Investigator, Simon Richards, Programme Leader Medical Ultrasound, Teesside University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AE14/11038; 14/NE/0023 (Other: Newcastle and North Tyneside 2 NRES committee)
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Sepsis; Severe Sepsis; Septic Shock
Keywords: Sepsis; ultrasound; inferior vena cava collapsibility
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm - Ultrasound (Other): All participants will have an Ultrasound measurement of their inferior vena cava at enrolment as described in the intervention
  Interventions: Other: Ultrasound of the inferior vena cava

INTERVENTIONS:
Other: Ultrasound of the inferior vena cava — B mode ultrasound of the inferior vena cava Measurements taken 2cm from the hepatic vein IVC junction or 3cm from the right atrium IVC junction

SUMMARY:
There is debate regarding the use of non invasive (ultrasound assessed) parameters of fluid volume status in patients with sepsis.

To establish the role of inferior vena cava ultrasound in guiding fluid resuscitation we first need to define the inferior vena cava collapsibility index in this population of patients.

The research question is: In adult patients with sepsis, severe sepsis and septic shock what is the mean baseline inferior vena cava collapsibility index (IVCCI) prior to fluid resuscitation.

DETAILED DESCRIPTION:
The study is an interventional cohort study using a convenience sample of adult patients in a university teaching hospital Emergency Department.

Eligible participants who consent to partake in the trial will have an ultrasound assessment of their inferior vena cava performed and the IVCCI will be calculated at enrolment.

Care will be provided in line with the published guidelines on sepsis management from the Surviving Sepsis Campaign and the College of Emergency Medicine.

A sample size calculation has been performed which indicates that 112 patient with severe sepsis or septic shock will need to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* signs and symptoms of infection with 2 or more SIRS criteria (pulse rate >90/min, Temp > 38 Celsius < 36 Celsius, Respiratory rate > 20 breaths per minute, or white cell count >12 or <4 x 10^9/L)

Exclusion Criteria:

* in relation to this episode of care: Prior cardio pulmonary resuscitation, acute myocardial infarction, trauma, pregnancy or patient requiring immediate surgery.
* Patients who have received more than 20ml/Kg of IV fluid in the pre hospital environment
* Patients with known tricuspid regurgitation, congestive heart failure or pulmonary hypertension
* Patients receiving palliative terminal supportive care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2014-07; Primary Completion 2014-12 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Mean baseline inferior vena cava collapsibility index | At enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Simon Richards, MHSc, Principal Investigator — Teesside University
Locations (1):
- St James's University Hospital, Leeds, West Yorkshire, United Kingdom